CLINICAL TRIAL: NCT02826135
Title: Study on Prediction of Fluid Responsiveness Using an Abdominal Compression-Induced Change of Blood Pressure in Children With Bidirectional Cavopulmonary Shunt or Fontan Pathway
Brief Title: Prediction of Fluid Responsiveness in Children With Single Ventricle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associated professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1603-156-752
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pediatric patients with hypovolemic state (Experimental): Right upper abdominal compression is performed in patients with hypovolemic signs including hypotension, decreased urine output or decreased central venous pressure. Changes of blood pressure during abdominal compression is continuously recorded.
  Interventions: Procedure: abdominal compression

INTERVENTIONS:
Procedure: abdominal compression — When there are clinical signs of hypovolemia, such as hypotension in pediatric patients with single ventricle, decreased urine output or decreased central venous pressure, right upper abdomen is gently compressed for 10 seconds. Changes of blood pressure are continuously recorded during this period. About 3 min later, intravenous colloid fluid 10 mL/kg is infused for 20 min.

SUMMARY:
The purpose of this study is to evaluate predictability of an abdominal compression-induced change of blood pressure for fluid responsiveness in children with single ventricle (bidirectional cavopulmonary shunt and Fontan tract).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate predictability of an abdominal compression-induced change of blood pressure for fluid responsiveness in children with single ventricle (bidirectional cavopulmonary shunt and Fontan tract).

When there are clinical signs of hypovolemia, such as hypotension, decreased urine output or decreased central venous pressure, right upper abdomen is gently compressed for 10 seconds. Changes of blood pressure are continuously recorded during this period. About 3 min later, intravenous colloid fluid 10 mL/kg is infused for 20 min.

To evaluate the change of cardiac output, transesophageal or transthoracic echocardiography is performed before and after fluid administration. In addition, hemodynamic parameters including pulse pressure variation, systolic pressure variation, pleth variability index and central venous pressure are also recorded before and after fluid administration.

Finally, patients will be divided into fluid responder group and non-responder group. If cardiac output measured using echocardiography increases over 15% after fluid administration, the patient is fluid responder. Using ROC curve, diagnostic power of abdominal compression-induced blood pressure change for fluid responsiveness will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing elective surgery, who require invasive blood pressure and central venous pressure monitoring during surgery
* Patients with bidirectional cavopulmonary shunt or fontan tract

Exclusion Criteria:

* renal, hepatic and pulmonary disease
* preoperative infection: increased CPR, WBC over 10,000, and with fever
* genetic and hematologic disease
* ventricular dysfunction
* increased intracranial pressure

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in stroke volume index after volume expansion | before and after fluid administration (20 min)

SECONDARY OUTCOMES:
Changes in pleth variability index after volume expansion | before and after fluid administration (20 min)
3.Changes in respiratory changes of peak aortic blood flow velocities after volume expansion | before and after fluid administration (20 min)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided